CLINICAL TRIAL: NCT03205878
Title: Improving Physical Activity in Obstructive Sleep Apnea Patients Treated With Continuous Positive Airway Pressure
Brief Title: Telecoaching to Improve Physical Activity in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S60283
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Physical Activity; Obstructive Sleep Apnea
MeSH Terms: conditions — Motor Activity; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients will receive standard care, being CPAP treatment
  Interventions: Device: CPAP
- Intervention group (Experimental): Patients will receive CPAP and telecoaching
  Interventions: Other: Telecoaching; Device: CPAP

INTERVENTIONS:
Other: Telecoaching — Patients in the intervention arm will receive a step counter and a cell phone with an app on which the amount of steps are daily sent to.
  Initial targets on steps per day will be discussed with the patient after an activity monitoring before the telecoaching procedure. Dependent whether the patient reaches his/her proposed goal each week, new goals are set.
  Arms: Intervention group
Device: CPAP — Patients will receive CPAP according to standard care

SUMMARY:
Patients with obstructive sleep apnea (OSA) are less physically active than healthy controls.

First choice of treatment for OSA is continuous positive airway pressure (CPAP) therapy with an improvement in oxygen saturation and sleep. No improvement on physical activity has been shown.

The current study would randomize patients in a standard care group (CPAP) and an intervention group (CPAP + telecoaching). Telecoaching will be performed for 3 months, with physical activity assessment before, after 3 months and 12 years.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 15 events/hour, measured by polysomnography
* < 7,500 steps per day
* Willing to start CPAP treatment
* Age between 18 and 65 years
* Signing the written informed consent

Exclusion Criteria:

* Patients with neuromuscular diseases
* Patients with chronic obstructive pulmonary disease and interstitial lung disease
* Patients with cardiac failure and ischemic heart failure
* Patients with comorbidities which could interfere with a normal biomechanical gait pattern and the possibility of increasing physical activity
* Patients with mental disability making it impossible to understand the study protocol and the use of electronic devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in steps per day after 3 months | The change will be measured after 3 months
  Steps per day as measured by a step counter

SECONDARY OUTCOMES:
The proportion of patients with an increase > 1,000 steps per day | After 3 months (end of telecoaching) and after 12 months
The proportion of patients with > 7500 steps/day | Before initiation of telecoaching (baseline), after 3 months (end of telecoaching) and after 12 months
Change in functional exercise capacity | 3 months and 12 months compared with baseline
  6-minute walking distance
Change in daytime sleepiness | 3 months and 12 months compared with baseline
  Epworth Sleepiness Scale
Change in sleep quality | 3 months and 12 months compared with baseline
  Pittsburgh Sleep Quality Index
Change in endothelial function | 3 months and 12 months compared with baseline
  Endo-PAT 2000 measurement
Change in body composition | 3 months and 12 months compared with baseline
  Bodystat 1500 measurement
Change in quality of life | 3 months and 12 months compared with baseline
  SF-36 questionnaire
Change in steps per day after 12 months | The change will be measured after 12 months
  Steps per day as measured by a step counter

IPD SHARING:
Plan to Share IPD: No